CLINICAL TRIAL: NCT03722706
Title: Improving Therapeutic Patient Education for Atopic Dermatitis: Evaluation of a Parent Handbook
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Jennifer LeBovidge, Attending Psychologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00029317
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Handbook (Experimental): handbook provided as an adjunct to standard AD management with a healthcare provider at BCH
  Interventions: Other: Educational handbook
- Control (No Intervention): standard management alone

INTERVENTIONS:
Other: Educational handbook — The intervention being evaluated in this study is an educational handbook for parents of children with atopic dermatitis (AD). The handbook was developed and written by the interdisciplinary study team (psychologist, allergist, nurse practitioner, dermatologists, primary care physician, dietitian). Content was based on practice guidelines for AD management, consensus recommendations for therapeutic patient education for AD, and clinical experience of our study team. Content includes topics central to effective AD management, such as pathophysiology/course, elements of treatment plans, and strategies to improve quality of life, such as breaking the itch-scratch cycle, improving sleep, and coping with social-emotional issues.
  Arms: Handbook

SUMMARY:
The objective of this research is to evaluate the effectiveness of an educational handbook for parents of children with atopic dermatitis (AD) in improving clinical outcomes for pediatric patients with AD and their parents. The handbook was developed by an interdisciplinary team of healthcare providers to facilitate therapeutic patient education as a routine component of care for pediatric patients with atopic dermatitis (AD). Patient education is an important element of practice management guidelines for AD, particularly given complex treatment plans and high rates of non-adherence in this population. Parents of children with AD will be randomized into either the handbook arm (handbook provided as an adjunct to standard AD management with a healthcare provider at Boston Children's Hospital) or the control arm (standard management alone). Participants will complete study measures at two time points: baseline (prior to a clinic visit appointment for AD care at Boston Children's Hospital), and 3-month follow-up. Data will be analyzed for change on study outcome measures (AD symptoms, AD severity, quality of life) and satisfaction with the handbook.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of atopic dermatitis
* Scheduled for clinic visit for evaluation/management of atopic dermatitis at Boston Children's Hospital

Exclusion Criteria:

* Parent is Spanish speaking
* Parent is foster parent

Ages: 30 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Patient-Oriented Eczema Measure (POEM) | baseline to 3-month follow-up
  parent-report of child's atopic dermatitis symptoms

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | baseline to 3-month follow-up
  healthcare provider-rating of atopic dermatitis severity
Infant's Dermatitis Quality of Life Index (IDQOL) | baseline to 3-month follow-up
  Quality of life associated with atopic dermatitis (for patients under 4 years)
Children's Dermatology Life Quality Index (CDLQI) | baseline to 3-month follow-up
  Quality of life associated with atopic dermatitis (for patients 4-16 years)
Dermatology Family Impact Questionnaire (DFI) | baseline to 3-month follow-up
  Parent quality of life associated with atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S LeBovidge, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No